CLINICAL TRIAL: NCT06689163
Title: An Open, Multicenter Phase Ib/II Study for the Treatment of Metastatic Prostate Cancer With HRS-1167 Tablets Combined With Abiraterone Acetate Tablets and Prednisone
Brief Title: A Study for the Treatment of Metastatic Prostate Cancer With HRS-1167 Tablets Combined With Abiraterone Acetate Tablets and Prednisone
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1167-201-A
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1167 combined with abiraterone acetate tablets (II) and prednisone (Experimental)
  Interventions: Drug: HRS-1167 tablets; Drug: Abiraterone Acetate tablets（II）; Drug: Prednisone Acetate tablets

INTERVENTIONS:
Drug: HRS-1167 tablets — HRS-1167 tablets
Drug: Abiraterone Acetate tablets（II） — Abiraterone Acetate tablets（II）
Drug: Prednisone Acetate tablets — Prednisone Acetate tablets

SUMMARY:
The purpose of this study was to observe and evaluate the tolerability, safety, and pharmacokinetics of HRS-1167 combined with abiraterone acetate tablets (II) and prednisone in patients with metastatic prostate cancer, determine the RP2D, and evaluate the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this study, signed informed consent, compliance is good, and are willing and able to comply with planned visits.
2. The age is above 18 years old, male.
3. Adenocarcinoma of the prostate confirmed with histologically or cytologically.
4. Metastatic lesions were confirmed by CT/MRI or radionuclide bone scan (99mTc).
5. ECOG score is 0 or 1.
6. An expected survival of ≥ 12 weeks.
7. Male subjects whose partner is women of childbearing potential (WOCBP) are required to use highly effective contraception from the date of signing the informed consent until 120 days after the last dose of the investigational drug.

Exclusion Criteria:

1. Received systemic antitumor therapy 4 weeks before starting study treatment; Participants who are participating in another clinical study or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or five half-lives of the investigational drug, whichever is shorter; Patients who had previously received anti-tumor proprietary Chinese medicine could be enrolled if the interval between the end of treatment and the first study was not less than 2 weeks.
2. Subjects had prior or co-existing malignancies , except for cured basal cell carcinoma of the skin, papillary carcinoma of the thyroid, and other malignancies that had been adequately treated and cured for ≥ 3 years prior to the first dose with evidence of no recurrence or metastasis.
3. Subjects had cancerous meningitis or untreated central nervous system metastases.
4. Imaging showed that the tumor invaded large blood vessels or had unclear boundary with blood vessels. Or patients whose tumors are judged by the investigators to be at high risk of invading vital blood vessels during treatment and causing fatal bleeding.
5. Patients with clinical symptoms of cancerous ascites and pleural effusion requiring puncture and drainage; Or received ascites, pleural effusion drainage within 14 days before the first dose.
6. Severe bone injury due to tumor bone metastasis, including poorly controlled severe bone pain, pathological bone fractures and spinal cord compression that occurred within the last 6 months or are likely to occur in the near future.
7. Pneumonia with past or current interstitial pneumonia/interstitial lung disease requiring treatment with the glucocorticoid system; Patients with active pneumonia or severe impairment of lung function confirmed by pulmonary function examination.
8. Systemic therapy with corticosteroids or other immunosuppressants within 2 weeks prior to the first dose.
9. Those with active pulmonary tuberculosis; Patients who had been adequately treated and had stopped anti-tuberculosis therapy for ≥3 months before the first dose could be enrolled.
10. Have high blood pressure that is not well controlled by antihypertensive medication; A history of hypertensive crisis or hypertensive encephalopathy.
11. Have clinical symptoms or diseases of the heart that are not well controlled.
12. Arterial/venous thrombosis events occurred within 6 months prior to the first dose.
13. Inability to swallow pills normally, or gastrointestinal dysfunction, may affect drug absorption.
14. Subjects who had a severe infection within 1 month prior to the first dose.
15. A known history of human immunodeficiency virus positive; Known to have active hepatitis.
16. The toxicity caused by previous antitumor therapy has not recovered to ≤ grade 1.
17. Live vaccine was administered within 4 weeks prior to the first dose or possibly using during the study.
18. In the judgment of the investigator, there are other factors that may affect the results of the study or cause the study to be terminated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days
Recommended phase II dose (RP2D) | 28 days
The dose suspension rate caused by drug-related adverse events | 2 years
The dose downregulation rate caused by drug-related adverse events | 2 years
The dose termination rate caused by drug-related adverse events | 2 years

SECONDARY OUTCOMES:
PSA response rate | 1 year
Time to PSA progression as assessed by the investigator | 1 year
Objective response rate (ORR) | 1 year
Disease control rate (DCR) | 1 year
Duration of response (DoR) | 1 year
Time to remission (TTR) | 1 year
Radiographic progression-free survival (rPFS) | 1 year
Overall survival (OS) | 3 years
Steady-state peak concentration (Cmax,ss) of HRS-1167 | 16 weeks
Adverse events | 2 years
12-lead electrocardiogram | 2 years
ECOG score | 2 years
Steady-state peak time (Tmax,ss) of HRS-1167 | 16 weeks
Steady-state valley concentration (Cmin,ss) | 16 weeks
Steady-state area under the concentration-time curve (AUCss) | 16 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided